CLINICAL TRIAL: NCT01552291
Title: The Impact of Preoperative Oral Glutamine Intake on the Immunocompetence and Outcomes of Malnourished Patients Undergoing Major Abdominal Surgery Due to Malignancies - A Randomized, Placebo-controlled Pilot Study
Brief Title: The Impact of Preoperative Oral Glutamine Intake on the Immunocompetence and Outcomes of Malnourished Patients Undergoing Major Abdominal Surgery Due to Malignancies
Acronym: Glutaminprojec
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 170/11
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Malnourishment; Gastrointestinal Tumors
Keywords: Malnourishment; Gastrointestinal tumors; Immunocompetence
MeSH Terms: conditions — Malnutrition; Digestive System Neoplasms | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamin (Active Comparator)
  Interventions: Dietary Supplement: Glutamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Glutamine — 30g oral glutamine / day for 5 days before surgery. Glutamine is an important nonessential amino acid and its intracellular concentration is much higher than that of other amino acids. Glutamine is released in large quantities from skeletal muscle and serves as an important carrier and donor of nitrogen
  Arms: Glutamin
Drug: Placebo — 30g oral maltodextrin / day for 5 days before surgery
  Arms: Placebo

SUMMARY:
Malnutrition occurs in up to 50% of patients requiring elective surgery for neoplastic diseases. It exerts a detrimental influence on outcome of surgery, because it can suppress immune function, exaggerate stress response and cause organ system dysfunction. Increased susceptibility to infection, protracted wound healing, impaired blood clotting and vessel wall fragility have been shown to be the leading causes of postoperative morbidity and mortality in malnourished patients undergoing major surgical resections.

This trial is designed as a prospective randomized, double-blinded, placebo-controlled pilot study in a academic single center in Switzerland. A total of 50 malnourished patients with gastro-intestinal tumors will receive orally glutamine or placebo-treatment during a period of 5 days prior to surgery. The investigators hypothesize that oral Glutamine administration is feasible, well tolerated, will decrease postoperative morbidity, will suppress postoperative cell damage and inflammatory response, and will improve the perioperative immunocompetence of the patients.

DETAILED DESCRIPTION:
Background

Malnutrition occurs in up to 50% of patients requiring elective surgery for neoplastic diseases. It exerts a detrimental influence on outcome of surgery, because it can suppress immune function, exaggerate stress response and cause organ system dysfunction. Increased susceptibility to infection, protracted wound healing, impaired blood clotting and vessel wall fragility have been shown to be the leading causes of postoperative morbidity and mortality in malnourished patients undergoing major surgical resections.

Immuno- or pharmaconutrition, defined as enteral or parenteral nutritional therapy based on a variety of products, such as omega-3-fatty acids, glutamine, arginine, sulfur-containing amino acids, nucleotides and anti-oxidants, is thought to have beneficial effects on postoperative recovery in a wide variety of surgical patients. Studies have shown its clinical effectiveness in terms of reduced postoperative complications, shortening the hospital stay and reduced hospitalization costs. Torosian et al. showed that severely malnourished patients benefit from preoperative nutrition, which reduce postoperative complications by 20%.

Although there is clinical evidence for the administration of immunonutrition to patients in the perioperative period, our understanding of the optimal type and time of immunonutrition, the characteristics of patients that benefit most, as well as the immunological mechanisms responsible for its beneficial effect is limited.

Objective

To assess in malnourished cancer patients the effect of 30g oral glutamine/day (3 sachets KABI® glutamine, Fresenius Kabi/day) for a preoperative course of 5 days on:

1. Postoperative morbidity (surgical site infections, pneumonia, sepsis, incidence of wound and fascial dehiscence, incisional hernia, anastomotic break down)
2. Nutritional status of the patients
3. Postoperative cell damage and inflammatory response
4. Perioperative immunocompetence

Methods

Seven days before surgery, the patients will receive a tetanus booster shot and will be randomly enrolled in either the 'glutamine group' or into the 'placebo group'. The patients as well as the responsible surgeons will be blinded.

* Patients in the 'glutamine group' will receive 30g oral glutamine / day for 5 days before surgery.
* Patients in the 'control group' will receive 30g oral maltodextrin / day for 5 days before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and surgically resectable carcinomas
* Candidates for elective surgery with an estimated surgical stress score
* A Nutritional Risk Screening 2002 (NRS-200232) score ≥3
* Age ≥ 18 years
* Completed primary immunization with tetanus toxoid
* Last tetanus booster ≥10 years back
* Informed consent

Exclusion Criteria

* Refusal to participate
* Clinically relevant alterations of the pulmonary renal of hepatic function
* Insulin-dependent diabetes mellitus
* Pre-existing autoimmune diseases and immune-deficiencies
* Neutropenia
* Pregnancy
* Age <18 years
* Last tetanus booster <10 years back
* Ongoing infection
* Intestinal obstruction at the time of entry into the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Morbidity | 6 weeks

SECONDARY OUTCOMES:
Postoperative cell damage | Up to seven days after surgery
Inflammatory response | Up to seven days after surgery
Nutritional status | Up to seven days after surgery
Perioperative immunocompetence | Seven and one day(s) before surgery. Postoperative week 1 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Beat Schnüriger, PD Dr. med., Principal Investigator — Department of visceral surgery and transplant surgery, Berne University Hospital
Locations (1):
- Department of visceral surgery and transplant surgery, Berne University Hospital, Bern, Switzerland